CLINICAL TRIAL: NCT04964076
Title: Clinical and Radiological Phenotypes of Patients With Stable COPD Between in Plateau and Plain
Brief Title: Clinical Phenotypes of COPD Patients Between in Plateau and Plain
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Tibet Autonomous Region People's Hospital (Other)
Responsible Party: Principal Investigator, Sun Yongchang, Peking University Third Hospital, Peking University Third Hospital
Other Study IDs: LM2020390
Record Dates: First submitted 2021-06-29; First posted 2021-07-15 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD patients in the plateau: We consecutively enrolled COPD patients visiting the outpatient of Respiratory Medicine at Tibet Autonomous Region People's Hospital from January 2018 to December 2021.
  Interventions: Other: No intervention
- COPD patients in the plain: We consecutively enrolled COPD patients visiting the outpatient of Respiratory Medicine at Peking University Third Hospital from January 2018 to December 2021.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
We aimed to collect clinical and radiological data of patients with stable COPD in plateau and plain, and compare the clinical phenotypic characteristics and imaging features of COPD patients in these two areas.

DETAILED DESCRIPTION:
The purpose of this study was to investigate the clinical phenotypic characteristics and imaging features of patients with stable chronic obstructive pulmonary disease (COPD) in plateau and plain. We conducted a cross-sectional study, collecting clinical data of stable patients in plateau and plain, and comparing the clinical phenotypic characteristics and imaging features of COPD patients in these two areas.

ELIGIBILITY:
Inclusion Criteria:

* meeting the diagnosis of COPD according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines and had definite airflow limitation with a post-bronchodilator forced expiratory volume in 1 second (FEV1) / forced vital capacity (FVC)<0.7.

Exclusion Criteria:

* age <40 years;
* subjects with airway diseases other than COPD;
* acute exacerbation of COPD in the past 3 months;
* active tuberculosis;
* cardiovascular or cerebrovascular events in the past 3 months;
* cognitive dysfunction such as vascular dementia or Alzheimer's disease;
* refusal to participate in this study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We consecutively enrolled patients with COPD from January 2018 to December 2021, who visited the outpatient of Department of Respiratory Medicine in Peking University Third Hospital or Tibet Autonomous Region People's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of respiratory symptoms | Data were obtained during the interview.
  COPD Assessment Test
Exacerbation | Data were obtained during the interview.
  Frequency of exacerbations in the past year
Spirometry testing | Data were obtained during the interview.
  FEV1 %predicted, FVC %predicted, ratio of FEV1/FVC
Emphysema | Within 3 months of the interview.
  The percentage of the LAA divided by total lung volumes (LAA%) was used as an index of the severity of emphysema in quantitative CT examination.
Airway remodeling -1 | Within 3 months of the interview.
  Bronchial wall thickness (WT, mm) was used as one of the measurements for assessment of airway remodeling in quantitative CT examination.
Airway remodeling -2 | Within 3 months of the interview.
  Luminal area (LA, mm2) was used as one of the measurements for assessment of airway remodeling in quantitative CT examination.
Airway remodeling -3 | Within 3 months of the interview.
  Bronchial wall area (WA, mm2) was used as one of the measurements for assessment of airway remodeling in quantitative CT examination.

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Sun, M.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China